CLINICAL TRIAL: NCT03297710
Title: Phase I Trial of TAS-102 and Concurrent Radiation Therapy for Patients With Locally Recurrent, Unresectable or Metastatic, Rectal Cancer
Brief Title: TAS-102 and Radiation Therapy in Treating Patients With Rectal Cancer That Is Locally Recurrent, Metastatic, or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1614; NCI-2017-01676 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1614 (Other: Mayo Clinic)
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-02

CONDITIONS: Rectal Adenocarcinoma; Recurrent Rectal Carcinoma; Stage IV Rectal Cancer AJCC v7; Stage IVA Rectal Cancer AJCC v7; Stage IVB Rectal Cancer AJCC v7
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Radiation; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TAS-102, radiation therapy) (Experimental): Patients receive trifluridine/tipiracil hydrochloride combination agent TAS-102 PO BID and undergo radiation therapy in 10 fractions on days 1-5 and 8-12 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102 — Given PO
  Other Names: Lonsurf; TAS-102; Trifluridine/Tipiracil

SUMMARY:
This phase I trial studies the side effects and best dose of trifluridine/tipiracil hydrochloride combination agent TAS-102 (TAS-102) when given together with radiation therapy in treating patients with rectal cancer that has come back, spread to other places in the body, or cannot be removed by surgery. Drugs used in chemotherapy, such as TAS-102, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving TAS-102 with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and dose-limiting toxicity of TAS-102 when administered in combination with concurrent radiation therapy in patients with locally recurrent or metastatic rectal cancer.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) to concurrent TAS-102 and radiation therapy in patients with locally recurrent or metastatic rectal cancer.

II. To determine the progression-free survival (PFS) in patients with locally recurrent or metastatic rectal cancer who receive concurrent TAS-102 and radiation therapy.

III. To determine the overall survival (OS) in patients with locally recurrent or metastatic rectal cancer who receive combined TAS-102 and radiation therapy.

IV. To determine quality of life (QoL) among patients with locally recurrent or metastatic rectal cancer who receive concurrent TAS-102 and radiation therapy.

V. To determine the number of patients who are able to undergo surgical resection following concurrent treatment with TAS-102 and radiation therapy. Of this subset of patients, the investigators will assess rates of pathologic complete response (pCR), tumor regression grade (TRG) and rates of R0 resection.

OUTLINE: This is a dose-escalation study of trifluridine/tipiracil hydrochloride combination agent TAS-102.

Patients receive trifluridine/tipiracil hydrochloride combination agent TAS-102 orally (PO) twice daily (BID) and undergo radiation therapy in 10 fractions on days 1-5 and 8-12 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4-6 weeks, and at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of locally recurrent or metastatic rectal adenocarcinoma

  * Note: Patients with locally recurrent/persistent disease within the pelvis after primary therapy (chemotherapy, surgery, and/or radiotherapy) are eligible
  * Note: Patients who have had prior pelvic radiotherapy with a total dose of =< 54 Gy are eligible
  * Note: Patients with or without metastatic disease (excluding untreated central nervous system [CNS] metastasis), with primary pelvic disease or pelvic recurrence are eligible
  * Note: Patients with pelvic disease that is potentially resectable or unresectable are eligible
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Expected life expectancy >= 12 weeks
* Obtained =< 14 days prior to registration: Absolute neutrophil count (ANC) >= 1500/mm^3
* Obtained =< 14 days prior to registration: Platelet count >= 100,000/mm^3
* Obtained =< 14 days prior to registration: Hemoglobin >= 9.0 g/dL
* Obtained =< 14 days prior to registration: Total bilirubin =< 1.5 x upper limit of normal (ULN) (in patients with well-documented Gilbert's syndrome and the total bilirubin is grade 1, then direct bilirubin value must be =< 1.0 mg/dL)
* Obtained =< 14 days prior to registration: Aspartate transaminase (AST) =< 2 x ULN (=< 5 x ULN for patients with liver involvement)
* Obtained =< 14 days prior to registration: Alanine aminotransferase (ALT) =< 2 x ULN (=< 5 x ULN for patients with liver involvement)
* Obtained =< 14 days prior to registration: Alkaline phosphatase =< 3 x ULN
* Obtained =< 14 days prior to registration: Creatinine =< 1.5 x ULN OR
* Obtained =< 14 days prior to registration: Calculated creatinine clearance must be >= 45 ml/min using the Cockcroft-Gault formula
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only; Note: patients must agree to adequate birth control during the study and for up to 6 months after discontinuation of study medication
* Patients must be able to take medications orally (i.e. no feeding tube)
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Able to complete questionnaires by themselves or with assistance

Exclusion Criteria:

* Primary resectable rectal cancer
* Prior treatment with TAS-102
* Chemotherapy or immunotherapy =< 28 days prior to registration
* Radiation therapy =< 28 days prior to registration; Note: patients with prior pelvic radiation therapy > 54 Gy are ineligible
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* Other concurrent chemotherapy, immunotherapy, or any ancillary antitumor therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Untreated CNS or leptomeningeal metastasis

  * Note: CNS or leptomeningeal disease must be stable for >= 3 months prior to registration
* History of seizure disorder
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Ascites, pleural effusion, or pericardial fluid requiring drainage in the last 4 weeks prior to registration
* Intestinal obstruction, uncontrolled gastrointestinal hemorrhage, pulmonary fibrosis, renal failure, liver failure, or cerebrovascular disorder
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or hepatitis B or C
* Patients with autoimmune disorders or history of organ transplantation who require immunosuppressive therapy
* History of myocardial infarction =< 12 months prior to registration, severe/unstable angina, systematic congestive heart failure (CHF) New York Heart Association classification III or IV or CHF requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Major surgery =< 4 weeks prior to registration (the surgical incision should be fully healed prior to drug administration or radiation therapy)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 28 days
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients.

OTHER OUTCOMES:
Best response as evaluated by the modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Best objective status recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started), assessed up to 6 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population.
Incidence and severity of adverse events graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 6 months
  Will be tabulated and summarized.
Incidence of toxicities graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 6 months
  Overall toxicity incidence as well as toxicity profiles by dose level and patient will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Median progression free survival | Up to 6 months
  Kaplan Meier curves will be utilized to estimate the median progression free survival in the expansion cohort.
Number of patients that make it to surgery | Up to 6 months
  Will assess rates of pathologic complete response (pCR), tumor regression grade (TRG), and rates of R0 resection.
Overall survival | Up to 6 months
  Kaplan Meier curves will be utilized to estimate the overall survival in the expansion cohort.
Quality of life (QoL) as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Up to 6 months
  Descriptive statistics of testing measures, including patients' pain and quality of life scores, will be calculated and correlated to treatment dose and response.
Time to progression | Up to 6 months
  Will be summarized descriptively.
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 6 months
  Will be summarized descriptively.
Time until any treatment related toxicity | Up to 6 months
  Will be summarized descriptively.
Time until hematologic nadirs (absolute neutrophil count [ANC], platelets, hemoglobin) | Up to 6 months
  Will be summarized descriptively.
Time until treatment related grade 3+ toxicity | Up to 6 months
  Will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Joleen Hubbard, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota